CLINICAL TRIAL: NCT05935241
Title: mHealth-Facilitated Physical Activity Toward Health (mPATH) Intervention for Low-Income Older Adults
Brief Title: mPATH for Low-income Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00396390; 1R01AG080613-01A1 (NIH)
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Sedentary Time; Insomnia; Cognitive Decline
Keywords: physical activity; memory; sleep
MeSH Terms: conditions — Sedentary Behavior; Sleep Initiation and Maintenance Disorders; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mPATH (Experimental): mPATH is a personalized physical activity intervention that includes personalized physical activity plans and training sessions, exercise at home by following personalized exercise videos, and biweekly phone coaching over 24 weeks, supported by wearable devices-enabled mHealth strategies. mHealth strategies and exercise videos will be used to support participant's physical activity during 6-12months
  Interventions: Behavioral: mPATH
- Education and Social control (Active Comparator): This attention control group is designed to match the intervention for mPATH's staff-subject interaction duration through monthly home visits in the first 6 months
  Interventions: Other: Attention Control

INTERVENTIONS:
Behavioral: mPATH — The active mPATH intervention takes 6 months including (1) The physical activity education session , (2)mHealth learning and practice; (3)Personalized physical activity training, plan, and biweekly phone calls over 24 weeks (4) mHealth strategies to encourage physical activity and facilitate intervention adherence (5) (5) mPATH during 6-12 months: mPATH will be delivered mainly in 24 weeks before the 6-month data collection. During 6-12 months, the participants will have access to study mHealth strategies, and exercise videos. No additional physical activity training by staff will be supported.
  Arms: mPATH
Other: Attention Control — A registered nurse from the study team will provide 6 monthly home visit (approximately 55-60 minutes each) to provide physical activity education, physical activity safety at home evaluation, feedback, and social activity (meaningful or enjoyable activities as identified by the participants, such as playing cards, doing arts and crafts, listening to music, talking about life history, etc.).
  Arms: Education and Social control

SUMMARY:
Although empirical research suggests that physical activity interventions benefit cognition and sleep in older adults in general, the possible benefit of physical activity is understudied in low-income older adults. The study aims to test the immediate and sustaining efficacy of an mHealth-facilitated Physical Activity Toward Health (mPATH) intervention on cognitive function and sleep in low-income older adults.

DETAILED DESCRIPTION:
Low-income older adults (LIOA) are a population at higher risk to develop Alzheimer's disease and related dementias (ADRD) and sleep disturbances. Although empirical research suggests that physical activity interventions benefit cognition and sleep in older adults in general, the possible benefit of physical activity is understudied in LIOA. The growing wearable device and mobile Health (mHealth) provide an innovative approach to deliver individually tailored physical activity interventions at home with flexible schedules to overcome barriers to physical activity in LIOA. In addition, limited research has examined if physical activity interventions impact the individual's Amyloid/Tau/ Neurodegeneration (ATN) Alzheimer's disease biological state and whether physical activity may promote cognition through impacting sleep and AD pathology. This randomized controlled trial is designed to examine the immediate and sustaining efficacy of an mHealth-facilitated Physical Activity Toward Health (mPATH) intervention on cognitive function and sleep in LIOA. mPATH is a personalized physical activity intervention that includes personalized physical activity plans and training sessions, exercise at home by following personalized exercise videos, and biweekly phone coaching over 24 weeks, supported by wearable devices-enabled mHealth strategies. mHealth strategies and exercise videos will be used to support participant's physical activity during 6-12months.

ELIGIBILITY:
Inclusion Criteria:

* self-reported difficulty of sleep
* lack of physical activity/exercise
* low household income
* capacity for moderate intensity exercise

Exclusion Criteria:

* untreated sleep apnea
* severe depression or anxiety
* dementia
* history of neurologic or psychiatric disorders, neurodevelopmental impairment, traumatic brain injury
* current enrollment in another clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in episodic memory as assessed by the Cogstate Alzheimer's Battery | Baseline, 6 months, 12 months
  Episodic memory will be measured by computerized cognitive batteries using the Cogstate Alzheimer's Battery.

SECONDARY OUTCOMES:
Change in Sleep efficiency as assessed by actigraphy | Baseline, 6 months, 12 months
  sleep efficiency will be measured by 7-day actigraph (reported as a percentage).

CONTACTS AND LOCATIONS:
Overall Officials: Junxin Li, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins University, School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
working on it
Supporting Information: Study Protocol, ICF, CSR
Time Frame: become available after the primary outcome paper published online
Access Criteria: with request